CLINICAL TRIAL: NCT00522002
Title: Connective Tissue Disease Leg Ulcer Etiology Study
Brief Title: CLUE Study: Connective Tissue Disease Leg Ulcer Etiology Study
Acronym: CLUE
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: American College of Rheumatology Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Victoria Shanmugam, Associate Professor of Medicine, George Washington University
Other Study IDs: IRB 2007-306
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Connective Tissue Diseases; Blood Coagulation Disorders; Leg Ulcers; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Systemic Scleroderma; Mixed Connective Tissue Disease
Keywords: Connective tissue diseases; Blood coagulation disorders; Leg ulcers; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Systemic Scleroderma; Mixed Connective Tissue Disease
MeSH Terms: conditions — Connective Tissue Diseases; Blood Coagulation Disorders; Leg Ulcer; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Mixed Connective Tissue Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To explore the hypothesis that leg ulcers are associated with hypercoagulable states, the CLUE study will evaluate patients with connective tissue disease associated leg ulcers, to identify risk factors (especially hypercoagulability and immunologic characteristics), characterize pathogenesis, predict response to therapy, and assess the impact of lower extremity ulcers on quality of life.

DETAILED DESCRIPTION:
Patients with non-healing leg ulcers who are over 18 years old will be eligible to enter the CLUE study. All eligible patients will be evaluated in both the Georgetown University Rheumatology Clinic and the Georgetown University Comprehensive Wound Healing Center. Since these evaluations are part of our routine care of patients, you need to have health insurance to be evaluated in our clinics.

WHAT DOES THE STUDY INVOLVE?

Enrollment in the CLUE study is voluntary, and will not affect your medical care at Georgetown University Hospital.

The standard evaluation of patients with non-healing leg ulcers evaluated in the Georgetown Division of Rheumatology includes an initial history and physical examination, along with hypercoagulable and autoimmune profiles. If this is your first visit to the rheumatology clinic the initial laboratory testing will require 3.5 tablespoons of blood. We will ask for your permission to review your medical record for previous blood test results so that you do not undergo unnecessary testing.

If you agree to participate in the CLUE study we will ask you to sign a consent form, allow us to photograph and measure your ulcers, and complete three brief pain and quality-of-life questionnaires.

If you continue to follow-up with the Georgetown Division of Rheumatology we will ask you to repeat these questionnaires at each clinic visit. If you prefer to follow-up elsewhere, we will ask for your permission to telephone you once per year to find out how your leg ulcers are doing.

WHAT TREATMENTS ARE AVAILABLE?

The CLUE Study is not a treatment trial. Treatment of your underlying connective tissue disease and leg ulcers will continue according to standard clinical care, as directed by doctors in the Division of Rheumatology and the Comprehensive Wound Healing Center.

In the future, studies testing new medications in patients with lower extremity ulcers may become available, and you may indicate on the consent form whether you would wish to be contacted regarding these studies.

WILL MY INFORMATION BE SECURE?

Information on CLUE study subjects will be stored on a password protected computer which will be kept in a locked room in the Division of Rheumatology. Your personal data will not be stored in this database and information will be identifiable only by a CLUE patient number.

WHAT ARE THE COSTS?

The CLUE Study is not a treatment trial. Just like any other doctors visit, you or your insurance will be charged for your initial evaluation and follow-up visits.

For more information on arranging an initial consultation in the Georgetown Division of Rheumatology, please call (202) 687-8233 and ask for an investigator to call you about the CLUE study.

Before your clinic visit can be scheduled, our staff will request that you have your primary care physician, rheumatologist or wound care specialist fax your previous medical records to our office at (202) 687-8579. If you have had previous scans, arteriograms or X-rays performed, please arrange to collect a copy of the scan and bring it to your appointment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory lower extremity ulcers
* Patients with Rheumatoid arthritis, Systemic Lupus Erythematosus, Systemic Scleroderma, Mixed Connective Tissue Disease or with lesions fulfilling a clinical diagnosis of Livedoid Vasculopathy

Exclusion Criteria:

* Lower extremity ulcers in the setting of diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory lower extremity ulcers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria K. Shanmugam, MD, Principal Investigator — Georgetown University Hospital; Thomas R. Cupps, MD, Study Chair — Georgetown University Hospital
Locations (1):
- Victoria Shanmugam, Washington D.C., District of Columbia, United States